CLINICAL TRIAL: NCT07080983
Title: Efficacy of Corneal Cross-Linking (CXL) in the Treatment of Pediatric Keratoconus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ehab Tharwat, Princibal Investigator, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pediatric Keratoconus
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cross-linking (Other)
  Interventions: Procedure: Crosslinking

INTERVENTIONS:
Procedure: Crosslinking — Corneal Cross-Linking (CXL) is a minimally invasive procedure used to strengthen the cornea by increasing the chemical bonds between collagen fibers. It is primarily used to treat keratoconus and corneal ectasia, conditions where the cornea becomes progressively thinner and weaker.

SUMMARY:
This prospective interventional study investigates the efficacy of corneal cross-linking (CXL) in managing progressive keratoconus in pediatric patients. The procedure involved standard epithelium-off CXL, and patients were followed to assess outcomes such as visual acuity, keratometric stability, and corneal thickness.

ELIGIBILITY:
Inclusion Criteria:

* Age between 8 and 18 years
* Clinical and topographic diagnosis of keratoconus based on the Belin/Ambrosio Enhanced Ectasia Display
* Evidence of progression within the past 6-12 months (e.g., an increase in maximum keratometry (Kmax) by ≥1.0 diopter, a decrease in minimal corneal thickness by ≥10 µm, or deterioration in visual acuity not attributable to other causes

Exclusion Criteria:

* Corneal scarring or opacities.
* Active ocular infection or inflammation.
* Prior ocular surgery or trauma.
* Autoimmune or connective tissue disorders.

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
keratometry (Kmax) | Baseline
  Kmax (Maximum Keratometry) is the steepest point of curvature on the cornea, and it is a key parameter in diagnosing and monitoring keratoconus.
keratometry (Kmax) | After 12 months
  Kmax (Maximum Keratometry) is the steepest point of curvature on the cornea, and it is a key parameter in diagnosing and monitoring keratoconus.
BCVA | Baseline
  Measurment of the visual acuity
BCVA | After 12 months
  Measurment of the visual acuity

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Ehab tharwat, Damietta, New Damietta
  - Al-Azhar university, Damietta

IPD SHARING:
Plan to Share IPD: Undecided